CLINICAL TRIAL: NCT02493608
Title: Scalpel vs Diathermy in Making Abdominal Wall Incision During Repeat Cesarean Delivery
Brief Title: Scalpel vs Diathermy in Repeat Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: L15-144
Record Dates: First submitted 2015-07-06; First posted 2015-07-09 (Estimated); Results first posted 2020-02-28 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Complications; Cesarean Section
MeSH Terms: interventions — Laser Therapy; Blade Implantation; Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- scalpel group (Active Comparator): Scalpel is the device used to make abdominal wall incision in this group of patient.
  Interventions: Device: scalpel
- Diathermy group (Active Comparator): In this study group, abdominal wall incisions are made with diathermy which is a electrosurgical instrument.
  Interventions: Device: Diathermy

INTERVENTIONS:
Device: scalpel — used to cut the abdominal wall.
  Other Names: Blade
  Arms: scalpel group
Device: Diathermy — Diathermy used to cut , coagulate the tissue
  Other Names: Bovie
  Arms: Diathermy group

SUMMARY:
The objective of this study is to compare scalpel vs. diathermy in abdominal wall incision in pregnant patients undergoing repeat elective cesarean delivery.

DETAILED DESCRIPTION:
It is hypothesized that wall incisions made by diathermy compared to scalpel during repeat cesarean delivery will have less incision time, as well as less blood loss. A second hypothesis is that the use of diathermy, compared with scalpel will not increase in post-operative pain.

1. This is a randomized prospective study in women undergoing elective repeat cesarean delivery at Medical Center Hospital in Odessa Texas.
2. Women undergoing cesarean delivery will be randomized into two groups: One group will undergo diathermy to incise the entire abdominal wall ,which includes skin, subcutaneous tissue, rectus muscle until the peritoneal cavity is visible. On the other group scalpel will be used to achieve the same aim.
3. A standardized abdominal wall incision will be made with either diathermy in cut mode or scalpel. Diathermy will be set in a cut mode with standard setting as per surgeons preference. All patients in the study will get standard skin incision in terms of length and depth which will be marked by a ruler.
4. Incision time ( measured in minutes and seconds with stop watch) and amount of bleeding will be measured. Blood loss will be calculated by weighing (in grams) the "used" lap sponges and comparing this to the weight (in grams0 of "fresh" lap sponges.
5. Post-operative pain will be measured by a Visual Analogue Scale (VAS). Measurements will be taken at 6:00 to 7:00 AM from post -op day 1 until hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Multiparous pregnant women 18 - 45 years.
* Gestational ages 37 weeks to 41 weeks,
* Undergoing repeat elective or repeat emergency cesarean deliveries.

Exclusion Criteria:

* Informed consent can't be obtained in a manner that allows for no impression of undue influence/pressure or sufficient time for patient to consider participation.
* Primary Cesarean deliveries - as these can bias the selection.
* Skin conditions such as infections, psoriasis, and eczema.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Caliendo, M.D, Principal Investigator — Texas Tech University
Locations (1):
- Medical Center Hospital, Odessa, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 were excluded from due to prior midline vertical skin incision.
Period: Overall Study
Arm/Group | Scalpel Group | Diathermy Group
Started | 48 | 48
Completed | 48 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Scalpel Group | Diathermy Group | Total
Number analyzed (Participants) | 48 | 48 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.9 (5.1) | 28.4 (5.3) | NA (NA) — Raw data is not available. PI has left institution.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 48 | 96
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Gravida [Mean (Standard Deviation); unit: Pregnancies] | 3.1 (1.1) | 3.5 (1.7) | NA (NA) — Raw data is not available. PI has left institution.
Para [Mean (Standard Deviation); unit: births] | 1.7 (0.8) | 1.7 (0.8) | NA (NA) — Raw data is not available. PI has left institution.
Weeks of Gestation [Mean (Standard Deviation); unit: Weeks] | 38.7 (0.7) | 38.4 (1.9) | NA (NA) — Raw data is not available. PI has left institution.
Height [Mean (Standard Deviation); unit: Centimeters] | 161.5 (7.5) | 160 (7.4) | NA (NA) — Raw data is not available. PI has left institution.
Weight [Mean (Standard Deviation); unit: kg] | 85.3 (17.9) | 86.9 (15.1) | NA (NA) — Raw data is not available. PI has left institution.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.7 (6.4) | 34.1 (5.7) | NA (NA) — Raw data is not available. PI has left institution.
Number of C-Sections [Mean (Standard Deviation); unit: number of C-sections] | 1.5 (0.7) | 1.7 (0.7) | NA (NA) — Raw data is not available. PI has left institution.
Type of Anesthesia [Count of Participants; unit: Participants]
  Spinal | 44 | 46 | 90
  Epidural | 4 | 2 | 6
Type of Surgery [Count of Participants; unit: Participants]
  Elective | 41 | 38 | 79
  Non-Elective | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: Incision Time .
Description: Time to make an abdominal wall incision from skin to rectus fascia.
Time Frame: during surgery
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Scalpel Group | Diathermy Group
Number analyzed (Participants) | 48 | 48
Seconds | 271.5 (109.31) | 188.17 (120.03)
Statistical Analysis 1: Comparison: Scalpel Group vs Diathermy Group; Test type: Other; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Post Operative Pain
Description: Done by VAS scale. Visual Analog Scale to measure pain. Scale range from 0 to 10 with higher values indicating worse pain.
Time Frame: Post Operative Day (POD) 1 and Day 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scalpel Group | Diathermy Group
Number analyzed (Participants) | 48 | 48
units on a scale
  POD 1 | 1.9 (2.6) | 2.6 (3.1)
  POD 2 | 3.2 (3.3) | 2.9 (3.2)
Statistical Analysis 1: Comparison: Scalpel Group vs Diathermy Group; Test type: Other; p = 0.218, t-test, 2 sided — POD 1
Statistical Analysis 2: Comparison: Scalpel Group vs Diathermy Group; Test type: Other; p = 0.638, t-test, 2 sided — POD 2

3. Secondary Outcome: Blood Loss
Description: Blood lost during incision/surgery
Time Frame: Blood lost during incision/surgery
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Scalpel Group | Diathermy Group
Number analyzed (Participants) | 48 | 48
grams | 15.98 (14.4) | 11.11 (15.43)
Statistical Analysis 1: Comparison: Scalpel Group vs Diathermy Group; Test type: Other; p = 0.113, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From surgery to discharge an average of two days.
Arm/Group | Scalpel Group | Diathermy Group
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 0/48 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-17): https://cdn.clinicaltrials.gov/large-docs/08/NCT02493608/Prot_SAP_000.pdf